CLINICAL TRIAL: NCT03287947
Title: LCI-GI-APX-NIN-001: Nintedanib in Metastatic Appendiceal Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low enrollment
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCI-GI-APX-NIN-001; 00021617 (Other: Advarra IRB)
Record Dates: First submitted 2017-07-31; First posted 2017-09-19 (Actual); Results first posted 2021-06-16 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-01

CONDITIONS: Appendix Cancer
MeSH Terms: conditions — Appendiceal Neoplasms | interventions — nintedanib

STUDY DESIGN:
Intervention Model Description: Single arm phase 2 study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- A (Experimental): Nintedanib
  Interventions: Drug: nintedanib

INTERVENTIONS:
Drug: nintedanib — Oral nintedanib, taken twice daily

SUMMARY:
The purpose of this trial is to evaluate the disease control rate of nintedanib in subjects with metastatic appendiceal cancer for whom initial fluoropyrimidine-based chemotherapy has failed. Based on previous studies, the anticancer activity of nintedanib in lung and ovarian cancer trials, along with the similarities between appendiceal and colorectal cancer and potentially ovarian cancer, warrant additional investigation for the optimal treatment of metastatic appendiceal carcinomas.

DETAILED DESCRIPTION:
The primary study objective is to evaluate the disease control rate. The secondary study objectives are to evaluate safety and toxicity, objective response rate, overall and 6-month progression free survival, and overall survival. Exploratory study objectives include evaluation of serum and ascites VEGF, hypertension, and paracentesis frequency in subjects with ascites at study entry.

ELIGIBILITY:
Inclusion Criteria

Subjects must meet all of the following criteria:

1. Age at least 18 years old
2. Histologically confirmed appendiceal carcinoma stage IV
3. Failure of initial fluoropyrimidine -based chemotherapy. Failure is defined as progression on or within 6 months of last day of therapy or intolerance of initial fluoropyrimidine-based chemotherapy.
4. Life expectancy at least 3 months
5. ECOG performance status score 0-2
6. Presence of measurable and/or evaluable, non-measurable disease according to RECIST 1.1 criteria
7. Written informed consent signed and dated by subject or Legally Authorized Representative (LAR) prior to admission to the study in accordance with ICH-GCP guidelines and to the local legislation.

Exclusion Criteria

Subjects must not meet any of the following criteria.

1. Prior treatment with nintedanib or any other VEGFR inhibitor
2. Known hypersensitivity to peanut or soya or to contrast media. History of hypersensitivity to contrast media is allowed if the subject is able to tolerate contrast media with pre-medication.
3. Chemo-, hormone-, radio-(except for brain and extremities) or immunotherapy, or therapy with monoclonal antibodies or small tyrosine kinase inhibitors within the past 4 weeks prior to treatment with the trial drug.
4. Radiotherapy to any target lesion within the past 3 months prior to baseline imaging when that target lesion is the only target lesion identified on baseline imaging, unless it has subsequently grown.
5. Persistence of clinically relevant therapy related toxicity from previous chemo and/or radiotherapy as determined by the investigator.
6. Active brain metastases (e.g. stable for <4 weeks, no adequate previous treatment with radiotherapy, symptomatic, requiring treatment with anti-convulsants; dexamethasone therapy will be allowed if administered as stable dose for at least one month) or leptomeningeal disease.
7. Radiographic evidence of cavitary or necrotic tumors.
8. Tumors with radiographic evidence (CT or MRI) of local invasion of major blood vessels.
9. Anti-neoplastic treatment for appendiceal cancer, with other investigational drugs or treatment in another clinical trial within 30 days before start of study treatment.
10. Therapeutic anticoagulation with drugs requiring INR monitoring (except low-dose heparin and/or heparin flush as needed for maintenance of an in-dwelling intravenous devise) or anti-platelet therapy (except for low-dose therapy with acetylsalicylic acid less than or equal to 325mg per day).
11. Major injuries and/or surgery within the past 4 weeks prior to start of study treatment, incomplete wound healing or planned surgery during the on-treatment study period.
12. History of clinically significant hemorrhagic or thromboembolic event in the past 6 months prior to consent.
13. Known inherited predisposition to bleeding or thrombosis.
14. Significant cardiovascular diseases (i.e. uncontrolled hypertension, unstable angina, history of infarction, congestive heart failure > NYHA II, serious cardiac arrhythmia, pericardial effusion) within the past 12 months prior to start of study treatment.
15. Proteinuria CTCAE grade 2 or greater.
16. Creatinine > 1.5x ULN or GFR < 45 ml/min.
17. Hepatic function: total bilirubin above normal limits; ALT or AST > 1.5x ULN in subjects without liver metastasis. For subjects with liver metastasis: total bilirubin above normal limits; ALT or AST > 2.5x ULN.
18. Coagulation parameters: International normalised ratio (INR) > 2x ULN, prothrombin time (PT) and partial thromboplastin time (PTT) > or equal to 1.5x ULN.
19. Absolute neutrophil count (ANC) < 1500/ml, platelets < 100000/ml, Hemoglobin < 9.0 g/dl.
20. Other malignancies at the time of signing the informed consent other than basal cell skin cancer or carcinoma in situ of the cervix.
21. Active serious infections if requiring systemic antibiotic or antimicrobial therapy.
22. Active or chronic hepatitis C and/or B infection.
23. Gastrointestinal disorders (like chronic diarrhea) or abnormalities that would interfere with absorption of the study drug. Subjects with this disorder may be allowed if able to tolerate anti-diarrheal medications like loperamide.
24. Serious illness or concomitant non-oncological disease such as neurologic, psychiatric, infectious disease or active ulcers (gastro-intestinal tract, skin) or laboratory abnormality that may increase the risk associated with study participation or study drug administration and in the judgment of the investigator would make the subject inappropriate for entry into the study.
25. Sexually active women of child-bearing potential and men who are sexually active with women of child-bearing potential and unwilling to use at least 2 medically acceptable methods of contraception (e.g. such as implants, injectables, combined oral contraceptives, some intrauterine devices or vasectomized partner for participating females, condoms for participating males) during the trial and for at least three months after end of active therapy. Female subjects will be considered of child-bearing potential unless surgically sterilized by hysterectomy or bilateral tubal/salpingectomy, or post-menopausal for at least 2 years.
26. Pregnancy or breast feeding; female participants of child-bearing potential must have a negative pregnancy test (B-HCG test in urine or serum) before commencing study treatment.

aa. Psychological, familial, sociological, or geographical factors potentially hampering compliance with the study protocol and follow-up schedule per the investigator.

bb. Alcohol or drug abuse which in the determination of the investigator would interfere with trial participation.

cc. Significant weight loss (> 10% of baseline weight) within past 2 months prior to consenting for the trial. Removal of ascites should not be calculated as weight loss.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-11-10 (Actual); Primary Completion 2019-09-03 (Actual); Study Completion 2019-10-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jimmy J Hwang, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Levine Cancer Institute, Charlotte, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Nintedanib: Participants received 200 mg oral nintedanib, taken twice daily.
Period: Overall Study
Arm/Group | Nintedanib
Started | 5 (Five subjects were enrolled to the study.)
Completed | 5 (All subjects enrolled discontinued treatment and are now off study.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Five subjects enrolled to the study at their initiations of nintedanib therapy.
Groups:
- Nintedanib: Subjects received 200 mg oral nintedanib, taken twice daily.
Arm/Group | Nintedanib
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.8 (15.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Ascites present at baseline [Count of Participants; unit: Participants] | 1

OUTCOME MEASURES:

1. Primary Outcome: Disease Control Rate
Description: The disease control rate is the proportion of those subjects with complete response, partial response, or stable disease, as defined by Response Evaluation Criteria in Solid Tumors Criteria (RECIST 1.1). Per RECIST 1.1 criteria for target lesions assessed by radiologic evaluation of CT and tumor measurements: Complete Response (CR), Disappearance of all target and non-target lesions, any pathological lymph nodes reduced in short axis to <10 mm; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), Neither sufficient shrinkage to qualify for PR nor PD; Disease Control Rate (DCR) = CR + PR + SD.
Time Frame: From first dose of study drug to date of progression as determined by RECIST 1.1, assessed up to 7.5 months.
Population: Subjects enrolled to the study at their initiations of nintedanib therapy and had measurable disease at baseline; four of five enrolled subjects had measurable disease at baseline.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Nintedanib
Number analyzed (Participants) | 4
Proportion of participants | .25 [.0064 to .8058]

2. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the duration from the start of nintedanib treatment to the date of death from any cause; subjects who are alive or lost to follow-up at the time of the analysis were censored at the last known date they were alive. Median overall survival was estimated using Kaplan-Meier methods. No formal comparative statistical analysis of overall survival was performed due to low accrual.
Time Frame: From date of first dose of study treatment to the date of death from any cause, assessed up to 14.5 months.
Population: All five enrolled subjects are evaluable for the analysis of overall survival.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nintedanib
Number analyzed (Participants) | 5
months | 2.62 [0.78 to 14.32]

3. Secondary Outcome: Progression-free Survival
Description: Progression-free survival was defined as the duration from the start of nintedanib treatment to the first occurrence of either progressive disease or death; disease progression was objectively determined per Response Evaluation Criteria in Solid Tumors Criteria (RECIST 1.1) or subjectively determined by the investigator. Per RECIST 1.1 criteria for target lesions assessed by radiologic evaluation of CT and tumor measurements: Progressive Disease (PD), >= 20% increase in the sum of the longest diameter of target lesions (at least 5 mm), or a measurable increase or progression in a non-target lesion, or the appearance of new lesions. Median progression-free survival was estimated using Kaplan-Meier methods. No formal comparative statistical analysis of progression-free survival was performed due to low accrual.
Time Frame: From date of first dose of study treatment to the date of progressive disease or death from any cause, whichever occurred first, assessed up to 7.5 months.
Population: All five enrolled subjects are evaluable for the analysis of progression-free survival.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nintedanib
Number analyzed (Participants) | 5
months | 1.34 [0.75 to 7.29]

4. Secondary Outcome: Treatment Administration of Nintedanib, as Measured by Average Daily Dose of Nintedanib.
Description: The average daily dose of nintedanib is calculated as the total cumulative dose (in mg) of nintedanib administered divided by the number of 28-day cycles on nintedanib treatment. Prescribed daily dose of nintedanib is 400 mg.
Time Frame: From the first dose of study drug to the last dose, assessed up to 7.5 months.
Population: Enrolled subjects returning bottles for drug accountability are included in the reporting of average daily dose of nintedanib.
Measure: Mean (Standard Deviation); unit: mg per cycle day
Arm/Group | Nintedanib
Number analyzed (Participants) | 3
mg per cycle day | 350.4 (48.4)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for subjects from enrollment until 30 days after last dose of study drug, assessed up to 8.5 months. All-Cause Mortality data was collected from enrollment until death, assessed up to 14.5 months.
Description: The attribution and severity of adverse events were classified and recorded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.
Arm/Group | Nintedanib
All-Cause Mortality (participants affected / at risk) | 5/5
Serious Adverse Events (participants affected / at risk) | 3/5
Other Adverse Events (participants affected / at risk) | 4/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nintedanib (N=5)
Death NOS (General disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Duodenal obstruction (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nintedanib (N=5)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Cardiac disorders - Other, Bradycardia (Cardiac disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Eye pain (Eye disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Localized edema (General disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (3)
Scalp pain (Skin and subcutaneous tissue disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-04-18): https://cdn.clinicaltrials.gov/large-docs/47/NCT03287947/Prot_SAP_000.pdf
  • Informed Consent Form (2017-10-20): https://cdn.clinicaltrials.gov/large-docs/47/NCT03287947/ICF_001.pdf